CLINICAL TRIAL: NCT01218711
Title: An Open Label, Randomized, 2-Period, 2-Treatment, Crossover, Single-Dose Bioequivalence Study of Fixed Dose Combination (FDC) of Losartan Potassium and Hydrochlorothiazide (100 mg / 25 mg Tablet) [Test Formulation, Torrent Pharmaceuticals Ltd., India] Versus Hyzaar® (100 mg / 25 mg Tablet) [Reference Formulation, Merck & Co., Inc., USA] in Healthy Human Volunteers Under Fasting Conditions.
Brief Title: Bioequivalence Study of Losartan Potassium and Hydrochlorothiazide (100 mg / 25 mg Tablet) [Test Formulation, Torrent Pharmaceuticals Ltd., India] Versus Hyzaar® (100 mg / 25 mg Tablet) [Reference Formulation, Merck & Co., Inc., USA] in Healthy Human Volunteers Under Fasting Conditions.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Other Study IDs: PK-07-067
Record Dates: First submitted 2010-10-07; First posted 2010-10-11 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Healthy
MeSH Terms: interventions — Losartan; Hydrochlorothiazide

INTERVENTIONS:
Drug: Losartan Potassium and Hydrochlorothiazide Tablets

SUMMARY:
Objective:

to compare the single dose bioavailability of Torrent's Losartan Potassium and Hydrochlorothiazide Tablets 1 × 100/25mg and Hyzaar® Tablets 1 × 100/25mg of Merck & Co., Inc.

Study Design:

Randomized, Two-Way Crossover, Single-Dose, Open-Label in 70 healthy human adult subjects

ELIGIBILITY:
Inclusion Criteria:

* The volunteers were excluded from the study based on the following criteria:

  * Sex: male.
  * Age: 18 - 45 years. .
  * Volunteer with BMI of 18-27 (inclusive both) kg/m2 with minimum of 50 kg weight.
  * Healthy and willing to participate in the study.
  * Volunteer willing to adhere to the protocol requirements and to provide written informed consent.
  * Non-smokers or smoker who smokes less than 10 cigarettes per day

Exclusion Criteria:

* The volunteers were excluded from the study based on the following criteria:

  * Clinically relevant abnormalities in the results of the laboratory screening evaluation.
  * Clinically significant abnormal ECG or Chest X-ray.
  * Systolic blood pressure less than 100 mm Hg or more than 140 mm Hg and diastolic blood pressure less than 60 mm Hg or more than 90 mm Hg.
  * Pulse rate less than 50/minute or more than 100/minute.
  * Oral temperature less than 95°P or more than 98.6°P.
  * Respiratory rate less than 12/minute or more than 20/minute
  * History of allergy to the test drug or any drug chemically similar to the drug under investigation.
  * History of alcohol or drug abuse
  * Positive breath alcohol test
  * Recent history of kidney or liver dysfunction.
  * History of consumption of prescribed medication since last 14 days or OTC medication since last 07 days before beginning of the study.
  * Volunteers suffering from any chronic illness such as arthritis, asthma etc.
  * History of heart failure.
  * HIV, HCV, HBsAg positive volunteers.
  * Opiate, tetra hydrocannabinol, amphetamine, barbiturates, benzodiazepines, Cocaine positive volunteers based on urine test.
  * Volunteers suffering from any psychiatric (acute or chronic) illness requiring medications.
  * Administration of any study drug in the period 0 to 3 months before entry to the study.
  * History of significant blood loss due to any reason, including blood donation in the past 3 months.
  * History of pre-existing bleeding disorder.
  * Existence of any surgical or medical condition, which, in the judgment of the chief investigator and/or clinical investigator/physician, might interfere with the absorption, distribution, metabolism or excretion of the drug or likely to compromise the safety of volunteers.
  * Inability to communicate or co-operate due to language problem, poor mental development or impaired cerebral function.

Ages: 18 Years to 45 Years | Sex: Male
Age Groups: Adult

PRIMARY OUTCOMES:
Bioequivalence based AUC parameters
Bioequivalence based on Cmax